CLINICAL TRIAL: NCT07088497
Title: Cmate Blood Glucose Analyzer: Clinical Comparison Study of Fasting Blood Glucose Levels in the Morning
Status: Completed | Type: Observational
Sponsor: Revlis Biotech Company Limited (Industry)
Collaborators: Taipei Medical University (Other); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202505166
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Glucose; Diabetes
Keywords: Non-invasive
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-diabetic subjects: 70 mg/dL< fasting blood glucose <100 mg/dL, HbA1c <5.7%
  Interventions: Behavioral: dietary control
- Pre-diabetic subjects: 100 mg/dL≤ fasting blood glucose <126 mg/dL, 5.7% ≤HbA1c<6.5%
  Interventions: Behavioral: dietary control
- Type 2 diabetes subjects: 126 mg/dL ≤ fasting blood glucose, 6.5% ≤HbA1c, no insulin injection
  Interventions: Behavioral: dietary control

INTERVENTIONS:
Behavioral: dietary control — Subjects are required to have dinner at a specific time on the night before the test and to remain fasting on the next day until the test.

SUMMARY:
As of February 2024, there are 529 million people worldwide living with diabetes. The number of diabetes patients continues to rise annually, and there is also a trend toward younger patients. Blood glucose management is crucial for prediabetes and diabetes patients. Effectively controlling blood glucose levels can reduce the risk of complications such as vascular complications, retinopathy, cardiovascular disease, and kidney disease. Traditionally, blood glucose monitoring in home settings has primarily relied on fingerstick whole blood samples combined with a blood glucose meter. However, this method poses risks associated with the disposal of used lancets and test strips, and the discomfort caused by the blood draw process can also lead to psychological stress for users. To enhance users' willingness to monitor blood glucose regularly and reduce environmental pollution from waste, the non-invasive blood glucose measurement system applied in this study is a non-invasive monitoring technology that is not a medical device and has not yet been marketed. It is currently undergoing the application process for FDA medical device certification in the United States. This trial will collect fasting venous plasma glucose levels, HbA1c, fingerstick whole blood glucose levels, and non-invasive glucose levels from patients in the morning. The primary analysis indicator is the correlation analysis between venous plasma glucose levels and non-invasive glucose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals willing to sign an informed consent form.
2. Adults aged 18 to 80 years.
3. Individuals with a past medical history diagnosed by a physician as meeting the following criteria, totaling 45 participants:

   A. Healthy participants (15 individuals): fasting blood glucose <100 mg/dL, HbA1c <5.7%.

   B. Pre-diabetic participants (15 individuals): fasting blood glucose ≤100 mg/dL and <126 mg/dL, HbA1c ≤5.7% and <6.5%.

   C. Patients with type 2 diabetes (15 individuals): fasting blood glucose ≥126 mg/dL, HbA1c ≥6.5%, and no insulin injection.
4. The proportion of males and females in each group is >30%.
5. Meets the signal acceptance criteria of the Cmate blood glucose analyzer.

Exclusion Criteria:

1. Individuals who refuse to sign the informed consent form.
2. Adults who lack legal capacity.
3. Individuals under the age of 18 or over the age of 80.
4. Individuals with a history of major cardiac conditions such as stroke, myocardial infarction, heart failure, coronary artery bypass surgery, stent placement, or pacemaker implantation.
5. Individuals with controlled heart disease who, during the screening visit, were found to have signal characteristics that cannot be used when screened with the Cmate blood glucose analyzer.
6. Type 1 diabetes patients.
7. Individuals with a history of gestational diabetes.
8. Pregnant women.
9. Individuals with fasting blood glucose levels below 70 mg/dL or above 200 mg/dL within the past three months.
10. Individuals whose signal characteristics do not meet the acceptance criteria of the Cmate blood glucose analyzer.
11. Individuals deemed ineligible for inclusion by the study principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are patients from Taipei Medical University Shuang Ho Hospital and nearby volunteers.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Non-invasive glucose levels accuracy | Within 60 days after the test day.
  Comparison of venous plasma glucose levels in test subjects with non-invasive glucose levels measured by the Cmate glucose analyzer.

SECONDARY OUTCOMES:
Non-invasive glucose levels accuracy | Within 60 days after the test day.
  Comparison of whole blood glucose levels measured at the fingertip of subjects with non-invasive glucose levels measured by the Cmate glucose analyzer.
HbA1c accuracy | Within 60 days after the test day.
  Comparison of venous plasma HbA1c levels of subjects with non-invasive HbA1c levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Chi Liu, Doctor, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Beginning 1 month after publication of results and ending at December 2026